CLINICAL TRIAL: NCT02285478
Title: Once Daily Darunavir/Ritonavir in HIV-infected Children 6-12 Years Old: a Pharmacokinetic Validation of Model Based Dosing Recommendations
Brief Title: Pharmacokinetics of Once Daily Darunavir/Ritonavir in HIV-infected Children
Acronym: DAPHNE
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AKF 13.03
Record Dates: First submitted 2014-10-27; First posted 2014-11-07 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Human Immunodeficiency Virus; Children
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Darunavir/ritonavir is one of the preferred antiretroviral agents as part of combination antiretroviral therapy for treatment of HIV-infected adults according to international guidelines. For children 3-12 years old, FDA has approved once daily dosing of darunavir/ritonavir. Dosing recommendations for children 6-12 years old have been approved based on a modelling and simulation procedure by the company.

This pharmacokinetic study is designed to validate the proposed dosing recommendation for once daily darunavir/ritonavir in HIV-infected children aged 6-12 years old.

DETAILED DESCRIPTION:
The EMA and FDA recommended weight band dosing for once daily DRV/r dosing in children 3 -12 years of age has been derived from pharmacokinetic modelling. Results from population pharmacokinetic modelling and simulation in these children predict similar DRV plasma exposures compared to treatment-naïve adults, but has not been formally studied in the target population. Although no clinical trial was conducted to collect exposure-safety data, the predicted exposures from the once daily dosing is supported by exposures observed in a paediatric clinical trial where twice-daily dosing was administered. To validate the weight band based dosing recommendations, we want to evaluate the pharmacokinetics of DRV/r administered once daily, using DRV tablets, in HIV-infected children.

Darunavir/ritonavir is one of the preferred antiretroviral agents as part of combination antiretroviral therapy for treatment of HIV-infected adults according to international guidelines. For children 3-12 years old, FDA has approved once daily dosing of darunavir/ritonavir. Dosing recommendations for children 6-12 years old have been approved based on a modelling and simulation procedure by the company.

This pharmacokinetic study is designed to validate the proposed dosing recommendation for once daily darunavir/ritonavir in HIV-infected children aged 6-12 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/carers are able and willing to sign the informed consent form prior to screening evaluations
2. Subject is HIV infected
3. Subject is at least 6 and less than 12 years at day of screening
4. Subject has a body weight of at least 15kg
5. Subject is able to swallow tablets
6. Subject has an undetectable viral load (<50 copies/mL) for the last 6 months prior to screening (at least 2 measurements)
7. ART regimen consists of darunavir/ritonavir and 2 NRTIs

Exclusion Criteria:

1. Inability to understand the nature and extent of the trial and the procedures required
2. Documented history of sensitivity/idiosyncrasy to darunavir or ritonavir medicinal products or its excipients
3. Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion
4. Abnormal renal or liver function (grade 3 or above)
5. Participation in a drug trial within 60 days prior to the first dose
6. Hemoglobin < 10 g/dL (6.0 mmol/L)
7. Children who have previously failed virologically on a PI containing regimen (where virological failure is defined as two successive HIV-1 RNA results >1,000 c/mL more than 24 weeks after starting cART, i.e. changes for toxicity or convenience are not counted as failure)
8. Acute illness
9. Receiving concomitant therapy except for prophylaxis for opportunistic infections; some treatments may be allowed, but must first be discussed with the principal investigator or project manager.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV-infected children (6-12 years) using once daily darunavir/ritonavir.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The exposure of darunavir, compared to the target exposure (AUC0-24) in adults | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Burger, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Result] Bastiaans DET, Geelen SPM, Visser EG, van der Flier M, Vermont CL, Colbers APH, Roukens M, Burger DM, van Rossum AMC; Dutch Paediatric HIV Study Group. Pharmacokinetics, Short-term Safety and Efficacy of the Approved Once-daily Darunavir/Ritonavir Dosing Regimen in HIV-infected Children. Pediatr Infect Dis J. 2018 Oct;37(10):1008-1010. doi: 10.1097/INF.0000000000001964. PMID 29474261